CLINICAL TRIAL: NCT00006010
Title: Phase II Trial of Gemcitabine and Docetaxel in Patients With Unresectable or Metastatic Hepatocellular Carcinoma
Brief Title: Gemcitabine Plus Docetaxel in Treating Patients With Unresectable or Metastatic Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0041; NCI-2012-02349 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000068019 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Liver Cancer
Keywords: localized unresectable adult primary liver cancer; advanced adult primary liver cancer; recurrent adult primary liver cancer; adult primary hepatocellular carcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Docetaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- docetaxel + gemcitabine (Experimental): Patients receive docetaxel IV over 15-60 minutes and gemcitabine IV over 30 minutes on days 1 and 8. Treatment repeats every 3 weeks. Patients achieving complete response after 2 courses of therapy receive 2 additional courses of therapy. Patients with stable disease or partial response continue therapy until disease progression.
  Patients are followed every 3 months for 1 year and then every 6 months for 4 years.
  Interventions: Drug: docetaxel; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: docetaxel
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one chemotherapy drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of gemcitabine plus docetaxel in treating patients who have unresectable or metastatic liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the six-month overall survival of patients with unresectable or metastatic hepatocellular carcinoma treated with gemcitabine and docetaxel.
* Determine tumor response and time to progression in this patient population treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Assess the pharmacokinetics of docetaxel in patients treated with this regimen.

OUTLINE: Patients receive docetaxel IV over 15-60 minutes and gemcitabine IV over 30 minutes on days 1 and 8. Treatment repeats every 3 weeks. Patients achieving complete response after 2 courses of therapy receive 2 additional courses of therapy. Patients with stable disease or partial response continue therapy until disease progression.

Patients are followed every 3 months for 1 year and then every 6 months for 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed unresectable or metastatic hepatocellular carcinoma not amenable to combined radiotherapy and chemotherapy or orthotopic liver transplantation
* Measurable disease, defined as at least 1 lesion that can be accurately measured in at least 1 dimension as at least 20 mm
* Evidence of disease progression by serial imaging or biochemical evidence of a rising alpha-fetoprotein by serial testing
* No history of brain or other CNS metastases not amenable to local therapy

  * Locally treatable CNS lesions (i.e., lesions treatable with surgery or radiosurgery) allowed if no evidence of CNS progression for at least 4 weeks after completion of therapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10.0 g/dL

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST no greater than 2.5 times ULN

Renal

* Creatinine no greater than 1.5 times ULN

Other

* No other malignancy within the past 5 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior hypersensitivity reaction to taxanes or other drugs formulated with polysorbate 80
* No grade 2 or greater peripheral neuropathy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 4 weeks since prior biologic therapy or immunotherapy
* No concurrent immunotherapy

Chemotherapy

* See Disease Characteristics
* Prior chemotherapy (excluding gemcitabine) for radiosensitization allowed
* At least 4 weeks since prior chemotherapy
* At least 6 months since prior chemoembolization
* No prior chemotherapy for metastatic disease
* No other concurrent chemotherapy

Endocrine therapy

* At least 4 weeks since prior hormonal therapy

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* No prior radiotherapy to 25% or more of bone marrow
* No concurrent radiotherapy

Surgery

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2001-09; Primary Completion 2004-05 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
six-month overall survival | at 6 months

SECONDARY OUTCOMES:
tumor response | Up to 5 years
time to progression | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven R. Alberts, MD, Study Chair — Mayo Clinic
Locations (17):
- United States (16):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Allan Blair Cancer Centre, Regina, Saskatchewan, Canada

REFERENCES:
- [Result] Alberts SR, Reid JM, Morlan BW, Farr GH Jr, Camoriano JK, Johnson DB, Enger JR, Seay TE, Kim GP. Gemcitabine and docetaxel for hepatocellular carcinoma: a phase II North Central Cancer Treatment Group clinical trial. Am J Clin Oncol. 2012 Oct;35(5):418-23. doi: 10.1097/COC.0b013e318219863b. PMID 21555932
- [Result] Kim GP, Alberts SR, Tschetter LK, et al.: Gemcitabine and docetaxel in patients with measurable unresectable or metastatic hepatocellular carcinoma (HCC), a North Central Cancer Treatment Group (NCCTG) phase II trial. [Abstract] J Clin Oncol 22 (Suppl 14): A-4270, 380s, 2004.